CLINICAL TRIAL: NCT05201274
Title: Effect of Baduanjin Sequential Therapy on the Cardiac Function and Exercise Endurance in Patients With AMI and Reduced Ejection Fraction After Primary PCI
Brief Title: Baduanjin Sequential Therapy and Cardiac Function of AMI With Reduced EF After PCI
Acronym: BST-AMI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenyang Northern Hospital (Other)
Responsible Party: Principal Investigator, Han Yaling, Director of cardiology, General Hospital of Northern Theater Command, Shenyang Northern Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BST-AMI
Record Dates: First submitted 2021-12-27; First posted 2022-01-21 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: AMI
Keywords: Acute myocardial infarction; Baduanjin; Percutaneous coronary intervention; Cardiac function; Physical function
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baduanjin sequential therapy (Experimental)
  Interventions: Behavioral: Baduanjin sequential therapy
- Aerobic exercise (Active Comparator)
  Interventions: Behavioral: Aerobic exercise

INTERVENTIONS:
Behavioral: Baduanjin sequential therapy — A detailed description of a standardized Baduanjin exercise protocol complied with the "Health Qigong Baduanjin Standard" enacted by the General Administration of Sports in 2003.
  Arms: Baduanjin sequential therapy
Behavioral: Aerobic exercise — Participants allocated to the usual exercise control group receive a closely supervised, group-format aerobic exercise program located at home or cardiac rehabilitation centre lasting 3 months. The program is consistent with the current recommended guidelines of moderate-intensity exercises for MI.
  Arms: Aerobic exercise

SUMMARY:
Acute myocardial infarction (AMI) is one of the leading causes of death around the world, with the potential for substantial morbidity and mortality. The increasing evidence indicates that exercise training has beneficial effects on LV remodelling in post-MI patients with greater benefits occurring when training earlier following MI, among which the earliest time for rehabilitation is one week after myocardial infarction. However, the effect of Baduanjin sequential therapy for patients after one week of AMI has yet to be assessed. Therefore, the aim of this study is to assess the impact of Baduanjin sequential therapy on cardiac and physical function in patients with AMI and reduced ejection fraction after primary PCI.

ELIGIBILITY:
Inclusion Criteria:

* Acute myocardial infarction undergoing primary percutaneous coronary intervention;
* Aged 18 years or over and under 80 years;
* 35% < LVEF < 50% and LV < 65mm;
* With informed consents

Exclusion Criteria:

* Severe symptomatic congestive heart failure (KILLIP cardiac function class III-IV);
* Malignant arrhythmias (ventricular fibrillation, ventricular tachycardia, frequent multiple source ventricular premature);
* Uncontrolled hypertension (systolic blood pressure greater than 160mmhg, diastolic blood pressure greater than 100mmhg);
* Life-threatening diseases with limited life expectancy <6 months;
* Inability or difficulty to exercise;
* Participation in other clinical trials

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-11-11 (Actual); Primary Completion 2023-02-11 (Estimated); Study Completion 2023-02-11 (Estimated)

PRIMARY OUTCOMES:
Left ventricular ejection fraction (LVEF) | baseline and 3 months
  The change in echocardiographic measures of left ventricular ejection fraction，(LVEF). LVEF in %.

SECONDARY OUTCOMES:
SF-36 | baseline and 3 months
  the SF-36 has 36 items grouped in 8 dimensions: physical functoning, physicial and emotional limitations, social functioning, bodily pain, general and mental health.
Generalized Anxiety Disorder 7-item (GAD-7) | baseline and 3 months
  The Generalized Anxiety Disorder 7 (GAD-7) is a 7-item instrument used to briefly measure or assess one of the most common mental disorders.
Patient Health Questionnaire (PHQ-9) | baseline and 3 months
  The PHQ-9 is the depression module, which scores each of the nine DSM-IV criteria as "0" (not at all) to "3" (nearly every day). It has been validated for use in primary care. It is not a screening tool for depression but it is used to monitor the severity of depression and response to treatment.
Seattle Angina Questionnaire (SAQ) | baseline and 3 months
  The Seattle Angina Questionnaire (SAQ), developed by Spertus and first reported in the literature in 1994, increasingly is being used to measure cardiac disease-specific quality of life in patients with CAD and
Minnesota Satisfaction Questionnaire (MSQ) | baseline and 3 months
  The Minnesota Satisfaction Questionnaire (MSQ) is initially designed to measure an employee's satisfaction with his or her job.
Traditional Chinese Medicine (TCM) symptom score scale | baseline and 3 months
  Traditional Chinese Medicine (TCM) symptom score scale is a score scale for evaluating patients' symptoms from the perspective of TCM. The full score is 30 points, 7-14 points are mild, 15-22 points are moderate and ≥23 points are severe.
CPET operators-Peak VO2/kg | baseline and 3 months
  Cardiopulmonary exercise testing ( CPET) is one kind of integrative evaluation of the subject's cardiopulmonary function under a certain exercise load. The information gathered during a CPET is used to calculate Peak VO2 (the highest level of oxygen consumption attained at peak exercise). (ml/kg/min)
CPET operators-metabolic equivalent (METs) | baseline and 3 months
  In cardiology, and especially when treadmill protocols are used, it is common to express the metabolic requirement for external work as the metabolic equivalent (MET). "MET" is defined as the equivalent of the resting metabolic oxygen requirement. One metabolic equivalent equals 3.5 ml/kg per minute. Exercise capacity (in METS) is a powerful predictor of mortality among men referred for exercise testing. (unit in METs)
CPET operators-peak O2-pulse | baseline and 3 months
  Another value calculated by CPET is the peak O2-pulse, which indicates how much blood one's heart can pump out with each beat (at the peak level of exercise). (ml/beat)
6-minute walk distance (6MWD) | baseline and 3 months
  A 6-minute walk test measures the distance patients can quickly walk in 6 minutes. (in meters)
Exercise compliance-exercise time | baseline and 3 months
  Exercise time. (in minutes)
Exercise compliance-Exercise frequency | baseline and 3 months
  Exercise frequency. (per week)
N-terminal pro-brain natriuretic peptide (NT-pro BNP) | baseline and 3 months
  N-terminal pro-brain natriuretic peptide (NT-pro BNP) in pg/ml
LV end-diastolic volume (LVEDV) | baseline and 3 months
  The change in echocardiographic measures of ventricular volumes (LV end-diastolic volume). LVEDV in ml.
LV end-systolic volume (LVESV) | baseline and 3 months
  The change in echocardiographic measures of ventricular volumes (LV end-systolic volume). LVESV in ml.

OTHER OUTCOMES:
The occurrence and composite of major adverse cardiac and cerebrovascular event (MACCE) | baseline and 3 months
  defined as recurrent myocardial infarction, any revascularization, readmission, stent thrombosis (ST) all-cause death and stroke)
Adverse events related to exercise rehabilitation | baseline and 3 months
  Adverse events related to exercise rehabilitation, such as fall.

CONTACTS AND LOCATIONS:
Overall Officials: Meili Liu, MD, Principal Investigator — General Hospital of Shenyang Military Region
Locations (1):
- General Hospital of Shenyang Military Region, Shenyang, Liaoning, China

REFERENCES:
- [Result] Perelshtein Brezinov O, Klempfner R, Zekry SB, Goldenberg I, Kuperstein R. Prognostic value of ejection fraction in patients admitted with acute coronary syndrome: A real world study. Medicine (Baltimore). 2017 Mar;96(9):e6226. doi: 10.1097/MD.0000000000006226. PMID 28248882
- [Result] Ibanez B, James S, Agewall S, Antunes MJ, Bucciarelli-Ducci C, Bueno H, Caforio ALP, Crea F, Goudevenos JA, Halvorsen S, Hindricks G, Kastrati A, Lenzen MJ, Prescott E, Roffi M, Valgimigli M, Varenhorst C, Vranckx P, Widimsky P; ESC Scientific Document Group. 2017 ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation: The Task Force for the management of acute myocardial infarction in patients presenting with ST-segment elevation of the European Society of Cardiology (ESC). Eur Heart J. 2018 Jan 7;39(2):119-177. doi: 10.1093/eurheartj/ehx393. No abstract available. PMID 28886621
- [Result] Yeh RW, Sidney S, Chandra M, Sorel M, Selby JV, Go AS. Population trends in the incidence and outcomes of acute myocardial infarction. N Engl J Med. 2010 Jun 10;362(23):2155-65. doi: 10.1056/NEJMoa0908610. PMID 20558366
- [Result] Haykowsky M, Scott J, Esch B, Schopflocher D, Myers J, Paterson I, Warburton D, Jones L, Clark AM. A meta-analysis of the effects of exercise training on left ventricular remodeling following myocardial infarction: start early and go longer for greatest exercise benefits on remodeling. Trials. 2011 Apr 4;12:92. doi: 10.1186/1745-6215-12-92. PMID 21463531